CLINICAL TRIAL: NCT07066722
Title: A Phase 1, Open-Label Study to Evaluate the Relative Bioavailability and the Effect of Food on VH4524184 Tablet Formulations, and to Evaluate the Potential for VH4524184 Drug-Drug-Interactions in Healthy Adult Participants
Brief Title: A Study to Evaluate VH4524184 Tablet Absorption, Effects of Food, and Interactions With Other Drugs in Healthy Adults
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 219890
Record Dates: First submitted 2025-07-03; First posted 2025-07-15 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: HIV Infections
Keywords: Drug-drug interaction; First-time in human; HIV; Bioavailability; Healthy Adult Participants
MeSH Terms: conditions — HIV Infections | interventions — Itraconazole; Rifabutin; Phenytoin; Metformin; Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Part 1A_VH4524184 (Sequence 1) (Experimental): Participants will receive VH4524184 tablet(s) of Dose level 1 followed by Dose level 2 in fasted condition.
  Interventions: Drug: VH4524184
- Part 1A_VH4524184 (Sequence 2) (Experimental): Participants will receive VH4524184 tablet(s) of Dose level 2 followed by Dose level 1 in fasted condition.
  Interventions: Drug: VH4524184
- Part 1A_VH4524184 (Sequence 3) (Experimental): Participants will receive VH4524184 tablet(s) of Dose level 3 followed by Dose level 2 in fasted condition.
  Interventions: Drug: VH4524184
- Part 1A_VH4524184 (Sequence 4) (Experimental): Participants will receive VH4524184 tablet(s) of Dose level 2 followed by Dose level 3 in fasted condition.
  Interventions: Drug: VH4524184
- Part 1B_VH4524184 (Sequence 5) (Experimental): Participants will receive VH4524184 tablet of Dose level 2 in fasted condition and then followed by intake of a high fat meal.
  Interventions: Drug: VH4524184
- Part 1B_VH4524184 Sequence 6) (Experimental): Participants will receive VH4524184 tablet of Dose level 2 following a high fat meal and then in fasted condition.
  Interventions: Drug: VH4524184
- Part 1B_VH4524184 (Sequence 7) (Experimental): Participants will receive VH4524184 tablet of Dose level 3 in fasted condition and then followed by intake of a high fat meal.
  Interventions: Drug: VH4524184
- Part 1B_VH4524184 (Sequence 8) (Experimental): Participants will receive VH4524184 tablet of Dose level 3 following a high fat meal and then in a fasted condition.
  Interventions: Drug: VH4524184
- Part 2_Cohort 1 (Experimental): Participants will receive VH4524184 tablet and Itraconazole.
  Interventions: Drug: VH4524184; Drug: Itraconazole
- Part 2_Cohort 2A (Experimental): Participants will receive VH4524184 and Rifabutin.
  Interventions: Drug: VH4524184; Drug: Rifabutin
- Part 2_Cohort 2B (Experimental): Participants will receive VH4524184 tablet and Phenytoin.
  Interventions: Drug: VH4524184; Drug: Phenytoin
- Part 2_ Cohort 3 (Experimental): Participants will receive Metformin, Digoxin and VH4524184 tablets.
  Interventions: Drug: VH4524184; Drug: Metformin; Drug: Digoxin

INTERVENTIONS:
Drug: VH4524184 — VH4524184 will be administered.
Drug: Itraconazole — Itraconazole will be administered.
  Other Names: Sporanox
  Arms: Part 2_Cohort 1
Drug: Rifabutin — Rifabutin will be administered.
  Other Names: Mycobutin
  Arms: Part 2_Cohort 2A
Drug: Phenytoin — Extended phenytoin sodium will be administered.
  Other Names: Dilantin
  Arms: Part 2_Cohort 2B
Drug: Metformin — Metformin will be administered.
  Other Names: Glumetza
  Arms: Part 2_ Cohort 3
Drug: Digoxin — Digoxin will be administered.
  Other Names: Lanoxin
  Arms: Part 2_ Cohort 3

SUMMARY:
The aim of the study is to gather information on how the drug behaves in healthy adults, how it is absorbed, and how it interacts when taken with other medicines.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be 18 to 60 years of age inclusive at the time of signing the Informed consent form (ICF).

2. Male or female

1. Male Participants: No restrictions for male participants
2. A female participant (female sex assigned at birth) is eligible to participate if she is not pregnant, or breastfeeding and the following condition applies: She is a woman of nonchildbearing potential (WONCBP).

   3. Participants who are overtly healthy as determined by medical evaluation 4. AST, ALT, alkaline phosphatase and bilirubin ≤ 1.5 x Upper Limit of Normal (ULN) 6. Capable of giving signed informed consent.

   Exclusion Criteria:
   1. History or presence of clinical conditions affecting drug absorption, metabolism, or elimination.,
   2. Pre-existing clinically relevant, gastro-intestinal pathology
   3. Abnormal glucose metabolism requiring insulin or medications.
   4. Clinically significant Abnormal blood pressure.
   5. History of Lymphoma, leukemia, or any malignancy within the past 5 years (3 years for resected basal or squamous epithelial carcinomas of skin).
   6. Breast cancer within the past 10 years.
   7. Current or chronic history of liver disease or known hepatic or biliary abnormalities.
   8. History of syncope, clinically significant palpitations, cardiac arrhythmias or cardiac disease or a family long QT syndrome.
   9. History of seizure(s) and / or other clinically significant neurological conditions.
   10. Pre-existing psychiatric condition, including depression, anxiety, and/or insomnia/sleep disturbances and / or suicidal ideation.
   11. History of drug hypersensitivity.

   13. Use of medications/supplements affecting cytochrome P450 enzymes within 7 to 14 days prior to dosing.

   14. Contraindications based on selected drug prescribing information. 15. Exposure to more than 4 new investigational products within 12 months 16. Current enrollment or past participation in another investigational study in which an investigational intervention was administered within the last 30 days.

   17. Estimated glomelular filtration rate (eGFR) < 90 mL/min or serum creatinine >1.1×ULN [Inker, 2021].

   18. Hemoglobin <12.5 g/dL for men and <11 g/dL for women. 19. Presence of Hepatitis B surface antigen (HBsAg) [and Hepatitis B core antibody (HBcAb)] at screening 20. Positive Hepatitis C antibody test result at screening 21. Positive SARS-CoV-2 test, having signs and symptoms which in the opinion of the investigator are suggestive of COVID-19.

   22.Positive pre- study drug/alcohol screen. 23. Poor metabolizers of CYP2C9 and / or CYP2C19 as assessed by genotype testing. HLA-B*1502 positive as applicable to specified cohort.

   Other exclusion criteria 24. Regular alcohol consumption exceeding specified limits. 25. Regular use of known drugs of abuse. 26. Nicotine use within 6 months. 27. Sensitivity or allergy to the study drug. 28. ALT >1.5×ULN. 29. Total bilirubin >1.5×ULN. 30. Significant arrhythmias or ECG findings that may compromise participant safety according to the investigator or VH Medical Monitor's assessment.

   31. For eligibility determination, triplicate ECGs are required. The criteria are:
   * Heart Rate: Excludes males with <45 or >100 bpm, females with <50 or >100 bpm.
   * PR Interval: Excludes any PR intervals <120 or >220 msec.
   * QRS Duration: Excludes durations <70 or >120 msec.
   * QTcF Interval: Excludes intervals >450 msec.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Part 1: Maximum plasma concentration (Cmax) for VH4524184 | Up to Day 18
Part 1: Area under the concentration-time curve from 0 to tau (AUC0-t) for VH4524184 | Up to day 18
Part 1: Area under the concentration-time curve from 0 to infinity (AUC0-inf) for VH4524184 | Up to day 18
Part 2: Cmax for VH4524184 | At Day 1, Day 14, Day 19 and Day 22
Part 2: AUC0-t of VH4524184 | At Day 1, Day 14, Day 19 and Day 22
Part 2: AUC0-inf of VH4524184 | At Day 1, Day 14, Day 19 and Day 22
Part 2: Cmax for metformin | At Day 1 and Day 15
Part 2: AUC0-t for metformin | At Day 1 and Day 15
Part 2: Cmax for Digoxin | At Day 1 and Day 15
Part 2: AUC0-t for Digoxin | At Day 1 and Day 15

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) and severity of AEs | From Day 1 up to Day 42
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. Severity of grades are defined as Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Potentially Life- Threatening.
Number of participants with AEs leading to discontinuation of study intervention | Throughout the study treatment period (from Day 1 up to Day 33)
Number of participants with Change in laboratory parameters | From Day 1 up to Day 42
Number of participants with maximum toxicity grade increase from baseline in laboratory parameters | From Day 1 up to Day 42
  Toxicity is graded using the DAIDS criteria Version 2.1 where grades were defined based on numeric criteria as follows Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: potentially life-threatening. A higher grade indicates greater severity.
Part 1: Time to maximum concentration (Tmax) of VH4524184 | At Day 1
Part 1: Apparent Terminal Half Life (T1/2) of VH4524184 | At Day 1
Part 1: Apparent oral clearance (CL/F) of VH4524184 | At Day 1
Part 2: Tmax of VH4524184 Following Single-Dose Administration with CYP3A4 Inhibitors and Inducers (Itraconazole, Rifabutin, Phenytoin) | At Day 1, Day 14, Day 19 and Day 22
Part 2: T1/2 of VH4524184 Following Single-Dose Administration with CYP3A4 Inhibitors and Inducers (Itraconazole, Rifabutin, Phenytoin) | At Day 1, Day 14, Day 19 and Day 22
Part 2: CL/F of VH4524184 Following Single-Dose Administration with CYP3A4 Inhibitors and Inducers (Itraconazole, Rifabutin, Phenytoin) | At Day 1, Day 14, Day 19 and Day 22
Part 2: Cmax for VH5424184 Following Comedication with Transporter Substrates with metformin and digoxin | At Day 1 and Day 15
Part 2: AUC0-t for VH5424184 Following Comedication with Transporter Substrates metformin and digoxin | At Day 1 and Day 15
Part 2: Cmax for Itraconazole Following Comedication with VH4524184 | At Day 1 and Day 14
Part 2: AUC0-t for Itraconazole Following Comedication with VH4524184 | At Day 1 and Day 14
Part 2: Cmax for Rifabutin Following Comedication with VH4524184 | At Day 1 and Day 11
Part 2: AUC0-t for Rifabutin Following Comedication with VH4524184 | At Day 1 and Day 19
Part 2: Cmax for Phenytoin Following Comedication with VH4524184 | Day 1 and Day 22
Part 2: AUC0-t for Phenytoin Following Comedication with VH4524184 | Day 1 and Day 22

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - GSK Investigational Site, Lenexa, Kansas
  - GSK Investigational Site, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.viiv-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.viiv-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf